CLINICAL TRIAL: NCT01099540
Title: Phase II Study of Pazopanib Monotherapy in Patients With Unresectable, Metastatic Neuroendocrine Tumor
Brief Title: Study of Pazopanib Monotherapy in Patients With Unresectable, Metastatic Neuroendocrine Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-09-090
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Neuroendocrine Tumor
Keywords: neuroendocrine tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental)
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 800 mg qd daily

SUMMARY:
To determine the response rate of pazopanib when administered as monotherapy in patients with unresectable neuroendocrine tumor.

ELIGIBILITY:
Inclusion Criteria:

* low to intermediate grade neuroendocrine tumor not amenable to surgery or local therapy

Exclusion Criteria:

* poorly differentiated (high grade or anaplastic)/small cell, pheochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
response rate | 1~2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Cancer Center, Seoul, South Korea

REFERENCES:
- [Derived] Ahn HK, Choi JY, Kim KM, Kim H, Choi SH, Park SH, Park JO, Lim HY, Kang WK, Lee J, Park YS. Phase II study of pazopanib monotherapy in metastatic gastroenteropancreatic neuroendocrine tumours. Br J Cancer. 2013 Sep 17;109(6):1414-9. doi: 10.1038/bjc.2013.470. Epub 2013 Aug 29. PMID 23989950